CLINICAL TRIAL: NCT00236795
Title: An Open-label Study to Evaluate the Contraceptive Efficacy and Safety of the Transdermal Contraceptive System of 17-deacetylnorgestimate and Ethinyl Estradiol With the Oral Contraceptive Triphasil.
Brief Title: A Study of Efficacy and Safety With the Transdermal Contraceptive System Versus Triphasil.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005506
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-11

CONDITIONS: Contraception; Female Contraception
Keywords: contraception; hormonal contraception; oral contraception; steroid, ethinyl estradiol, horgestimate, levonorgestrel contraception; transdermal.
MeSH Terms: interventions — norelgestromin; Ethinyl Estradiol; Ethinyl Estradiol-Norgestrel Combination

INTERVENTIONS:
Drug: norelgestromin + ethinyl estradiol; triphasil.

SUMMARY:
The purpose of the study was to compare the contraceptive efficacy and safety of the transdermal patch to Triphasil.

DETAILED DESCRIPTION:
This is an open-label, multicenter, worldwide study to evaluate the contraceptive efficacy, safety, cycle control, compliance, and subject satisfaction of the transdermal patch compared with Triphasil. Fourteen hundred healthy women will receive study medication for either 6 or 13 cycles. The first 33% of subjects (~265 transdermal patch subjects and 200 Triphasil subjects) will be expected to complete 13 cycles of medication. All subsequent subjects will be expected to complete 6 cycles. The ratio of subjects assigned to the transdermal patch arm of the study and to the Triphasil arm will be 4:3. At admission (Visit 1) study drug (plus 3 reserve patches), diary cards and subject instructions for Cycle 1 are dispensed. The first patch will be applied and Triphasil pill will be taken on the first day of menses. Study medication and diary cards will be issued on day 28 of Cycles 1 (Visit 2) and 3 (Visit 3), and those continuing for 13 cycles will receive study drug again (plus 3 reserve patches) on day 28 of Cycles 6 (Visit 4) and 9 (Visit 5). Diary cards and empty medication packages will be collected at every visit. Final visits are on day 28 of Cycles 6 and 9. Diary card information is used to record compliance and bleeding information (to assess cycle control). Contraceptive efficacy was assessed by means of the Pearl Index and life table analysis (gross cumulative probability of pregnancy). Safety evaluations were based on adverse events, which were collected throughout the study, and changes in physical examinations, gynecologic examinations, vital signs, and laboratory results from prestudy to final visit. A transdermal patch, containing 6 mg NGM and 0.75 mg EE, delivering 250 ug NGM and 25 ug EE over 24 hours for 7 days, is worn for 1 week and replaced for 3 consecutive weeks.The fourth week is patch-free. A Triphasil pill is taken for 28 consecutive days at the same time each day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, nonpregnant women with regular menstrual cycles
* sexually active and at risk of pregnancy
* acceptable body mass index (BMI)
* last term pregnancy at least 42 days prior, nonlactating, with 1 normal menstrual cycle since
* sitting BP<140mmHg/<90mmHg
* 1 normal menstrual cycle since removal of IUD or norplant
* agreement to use study drug for contraception for up to 13 cycles, except when backup contraception is required for disease protection or patch detachment
* agree not to use other systemic steroid medication

Exclusion Criteria:

* Presence, history, hereditary predisposition or risk of deep vein thrombophlebitis or thromboembolic disorders
* cerebral vascular or coronary artery disease, hypertension, or severe migraines
* liver tumor resulting from estrogen-containing products
* diabetes mellitus
* cholestatic jaundice, liver or renal disease
* abnormal PAP smear
* undiagnosed abnormal vaginal bleeding
* thyroid disorder
* dermal hypersensitivity
* carcinoma of breast, genital tract or other estrogen-dependent neoplasia
* received any depot hormone injection within prior 6 months
* smoking women over 35 years of age.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1494 (Actual)
Dates: Start 1997-01; Study Completion 1999-03 (Actual)

PRIMARY OUTCOMES:
Contraceptive efficacy of the 2 treatments was estimated by determination of pregnancy rates, using the Pearl Index and life table analysis (cumulative probability of pregnancy). Safety was evaluated throughout the study.

SECONDARY OUTCOMES:
Cycle control and compliance were assessed with diary cards containing bleeding and dosing information.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Zieman M, Guillebaud J, Weisberg E, Shangold GA, Fisher AC, Creasy GW. Contraceptive efficacy and cycle control with the Ortho Evra/Evra transdermal system: the analysis of pooled data. Fertil Steril. 2002 Feb;77(2 Suppl 2):S13-8. doi: 10.1016/s0015-0282(01)03275-7. PMID 11849631
- [Result] Zacur HA, Hedon B, Mansour D, Shangold GA, Fisher AC, Creasy GW. Integrated summary of Ortho Evra/Evra contraceptive patch adhesion in varied climates and conditions. Fertil Steril. 2002 Feb;77(2 Suppl 2):S32-5. doi: 10.1016/s0015-0282(01)03262-9. PMID 11849634
- See also: A study of efficacy and safety with the transdermal contraceptive system versus Triphasil. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=661&filename=CR005506_CSR.pdf